CLINICAL TRIAL: NCT00418652
Title: Interruption of Dorsal Visual Stream Using TMS in Normal Controls
Brief Title: Interruption of Dorsal Visual Stream Using TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Amiaz Revital, MD - Senior Psychiatrist, Sheba Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHEBA-06-4252-RA-CTIL
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: Normal Controls

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- No TMS stimulation (No Intervention): The patients performed 2 tasks: a study and a control assignments with no TMS stimulation.
  Interventions: Device: No TMS intervention
- TMS over the dorsal stream (Experimental): The patients performed 2 tasks: a study and a control assignments under TMS stimulation over the dorsal stream area (PO3 EEG site).
  Interventions: Device: TMS over the PO3 EEG site
- TMS over the vertex (Sham Comparator): The patients performed 2 tasks: a study and a control assignments under TMS stimulation over the vertex area.
  Interventions: Device: TMS over the vertex

INTERVENTIONS:
Device: No TMS intervention — In the "no TMS" condition, no simulation was given and no coil placed near participants' heads.
  Arms: No TMS stimulation
Device: TMS over the PO3 EEG site — 10Hz TMS over the dorsal stream (PO3 EEG site)
  Other Names: MAGSTIM biphasic stimulator
  Arms: TMS over the dorsal stream
Device: TMS over the vertex — 10Hz TMS for over vertex.
  Other Names: MAGSTIM biphasic stimulator
  Arms: TMS over the vertex

SUMMARY:
Trans Cranial Magnetic Stimulation (TMS) over dorsal visual system will disturb the ability to identify objects with decreased level of fragmentation

DETAILED DESCRIPTION:
The participants performed two tasks under three different TMS conditions: no TMS, 10Hz TMS for over the dorsal stream (PO3 EEG site) or over the vertex.

First they performed a perceptual closure task which asked them to identify an object in a series of six progressively less degraded pictures.

Then, they also performed a control task previously shown not to be mediated by the LOC and not to be impaired in schizophrenia: The perception of illusory contours.

ELIGIBILITY:
Inclusion Criteria:

* Normal controls

Exclusion Criteria:

* neurological, ophthalmological or psychiatric problems
* family history of schizophrenia
* left handed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-01; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Results of the study assignments performed by the participants during the study. | The participants performed the tasks once during their study visit
  The subjects performed 2 tasks:
  The primary dependent measures consisted of the level of detail needed for correct object identification, response accuracy, and response time in milliseconds for correct responses.
  Illusory Contour Task: Subjects also performed a pulsed pedestal task, Participants were shown 55 drawings for 500 ms each. Some drawings contained partial contours which defined a geometric shape, while in others the contours did not define a shape. Participants were asked to indicate whether they recognized a geometric shape or not. Accuracy and response time were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Revital Amiaz, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Psychiatry Clinic - Sheba Medical Center, Tel Litwinsky, Israel